CLINICAL TRIAL: NCT02036983
Title: Comparison of an Ultrasound Guided Bilateral Transversus Abdominis Plane Block With Dexamethasone and Preperitoneal Instillation of Local Anesthetic With Dexamethasone to a Standard Anesthetic Technique for Analgesic Efficacy and Patient Satisfaction Following a Total Extraperitoneal Bilateral Inguinal Hernia Repair: A Prospective Randomized Single Blinded Study
Brief Title: Comparison of a Bilateral TAP Block and Preperitoneal Instillation of Local Anesthetic for a Total Extraperitoneal (TEP) Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1308124192
Record Dates: First submitted 2013-12-05; First posted 2014-01-15 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-08

CONDITIONS: Bilateral Inguinal Hernia Repair
Keywords: Ultrasound guided; Bilateral Transversus abdominis Plane Block; Dexamethasone; Preperitoneal Instillation; Local Analgesic; Efficacy; Total Extraperitoneal Bilateral Inguinal hernia repair
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ultrasound guided bilateral TAP block (Active Comparator): Ultrasound guided TAP Block with local anesthetic and dexamethasone.
  Interventions: Procedure: Transversus abdominis plane block (TAP BLOCK)
- Instillation of surgical site with local anesthestic. (Active Comparator): Instillation of surgical site under direct visualization with local anesthetics and dexamethasone.
  Interventions: Procedure: Instillation of surgical site with local anesthetic.
- Control Group (Placebo Comparator): Standard anesthetic technique
  Interventions: Procedure: Opioid IV medications (Control)

INTERVENTIONS:
Procedure: Transversus abdominis plane block (TAP BLOCK) — Ultrasound guided TAP block with local anesthetics and dexamethasone.
  Arms: Ultrasound guided bilateral TAP block
Procedure: Instillation of surgical site with local anesthetic. — Instillation of surgical site with local anesthetics and dexamethasone.
  Arms: Instillation of surgical site with local anesthestic.
Procedure: Opioid IV medications (Control) — Standard anesthetic technique.
  Arms: Control Group

SUMMARY:
Comparison of an ultrasound guided bilateral TAP (transversus abdominis plane) block with dexamethasone and preperitoneal instillation of local anesthetic with dexamethasone under direct visualization will be compared it to a standard anesthetic technique (control) following a TEP (total extraperitoneal) bilateral hernia repair. The investigators are hypothesizing that the bilateral TAP block and preperitoneal instillation of local anesthetics with the addition of dexamethasone are superior in terms of patient satisfaction and post-operative pain control when compared to a standard anesthetic technique (no regional technique).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 yrs of age
* American Society of Anesthesiologists (ASA) physical status 1-3
* Scheduled for outpatient TEP bilateral inguinal hernia repair

Exclusion Criteria:

* Patients refusal to participate
* inability to give consent
* drug allergies to medications used in study
* pregnancy
* bleeding diathesis
* conversion to an open procedure
* any subject whose anatomy, or surgical procedure, in the opinion of the investigator might preclude the potential successful performance of a TAP block
* any subject whose anatomy, or surgical procedure, in the opinion of the investigator, might preclude the potential successful performance of a TAP block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (Day 1)
  Assessment will be done postoperatively using a Quality of Recovery 40 (QoR-40) questionnaire after surgery.

SECONDARY OUTCOMES:
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (Day 0 to 1)
  Total opioid use in the post anesthesia care unit (PACU) and the period following surgery.
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (day 0)
  Pain scores in the PACU
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (day 1)
  Pain scores post-operatively.
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (day 0 to 1)
  Any side effects secondary to any of the post-operative pain procedures.
Assess the efficacy of a bilateral TAP block and preperitoneal instillation of local anesthetic to a standard anesthetic technique for TEP hernia repair | Post-operatively (day 0)
  Time spent in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Sakamoto, M.D., Principal Investigator — Indiana University
Locations (1):
- Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Sakamoto B, Harker G, Eppstein AC, Gwirtz K. Efficacy of Local Anesthetic With Dexamethasone on the Quality of Recovery Following Total Extraperitoneal Bilateral Inguinal Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2016 Dec 1;151(12):1108-1114. doi: 10.1001/jamasurg.2016.2905. PMID 27653293